CLINICAL TRIAL: NCT04318418
Title: ACE Inhibitors, Angiotensin II Type-I Receptor Blockers and Severity of COVID-19
Acronym: CODIV-ACE
Status: Completed | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Augusto Di Castelnuovo, MSc, PhD, Neuromed IRCCS
Other Study IDs: DEP_012020
Record Dates: First submitted 2020-03-19; First posted 2020-03-24 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: COVID-19
Keywords: Angiotensin receptor-blocker and ACE inhibitors drugs
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients who developed severe COVID-19 disease (including fatal events)
- Controls: Infected patients who did not develop severe COVID-19 respiratory disease (including individuals who recovered from the infection)

SUMMARY:
Hypothesis Very recent evidences supports the hypothesis that the novel coronavirus 2019 (2019-nCoV) uses the SARS-1 (severe acute respiratory syndrome

) coronavirus receptor angiotensin converting enzyme 2 (ACE2) for entry into target cells. The epidemiological association between Angiotensin receptor-blocker (ARB) or ACE inhibitors (ACE-I) use and severe sequelae of 2109-nCoV infection disease COVID-19 has not been yet conclusively demonstrated, but may have important consequences for population health.

Aim To retrospectively test whether 2019-nCoV patients treated with ACE-I or ARB, in comparison with patients who not, are at higher risk of having severe COVID-19 (including death).

Population Hospitalized patients with confirmed COVID-19 infection (any type).

Study design Patients will be divided in two groups, a) controls: individuals who did not develop severe COVID-19 respiratory disease (including individuals who recovered from the infection) and b) cases: individuals who developed severe COVID-19 disease (including fatal events). Treatment with ACE-I or ARB, together with possible confounding will be assessed retrospectively.

Exposure Treatment for ACE-I or ARB.

DETAILED DESCRIPTION:
Background Very recent evidences support the hypothesis that the novel coronavirus 2019 (2019-nCoV) uses the SARS-1 coronavirus receptor ACE2 for gains entry into target cells. Angiotensin receptor-blocker (ARB) drugs, one of the most commonly used antihypertensive drug, typically increase ACE2 expression, often very markedly. With SARS-CoV-2 infection increased ACE2 expression very definitely would not be beneficial, and could be adverse. However, augmented ACE2 expression with ARB has been demonstrated in the kidneys and heart but has not been tested in the lungs. So, the hypothesis that using of ARB or ACE inhibitors (ACE-I) drugs during the COVID-19 may possibly be harmful is urgently to be verified in epidemiological studies.

Aim To retrospectively test whether 2019-nCoV patients treated with ARB or ACE-I, in comparison with patients who not, are at higher risk of having severe COVID-19 (coronavirus infection disease 2019), including death.

Population Hospitalized patients with confirmed COVID-19 infection (any type).

Outcome The project will retrospectively collect data on the most severe manifestation of COVID-19 occurred in 2019-nCoV infected patients during hospitalization. Severity will be classified as: hospital discharge with healing, asymptomatic, mild complications but not pneumonia, not severe pneumonia, severe pneumonia, acute respiratory distress syndrome (ARDS) and death. Classification of pneumonia will follow WHO (World Health Organization) criteria. Data on severity will be obtained from medical record at one-point time (at the moment of inclusion in the study).

Exposure Treatment for ARB or ACE-I. When available, type of drugs will be recorded.

Study design Patients will be divided in two groups, a) controls: individuals who did not develop severe COVID-19 respiratory disease (including individuals who recovered from the infection) and b) cases: individuals who developed severe COVID-19 disease (including fatal events). Association between use of ACE-I or ARB and severity of COVID-19 will be assessed by using of multivariable logistic regression analysis. Data on potential confounders will be obtained by medical records: age, sex, time intervals from hospital admission to worse manifestation of COVID-19 and to eventual death or recovering, smoking, body mass index, history of myocardial infarction, diabetes, hypertension, cancer, respiratory disease, other morbidities, creatinine, insulin, glomerular filtration rate together with use of Tocilizumab, anti-aldosterone agents, diuretics, Kaletra, cortisone, Remdesivir, Hydroxychloroquine, Sacubitril or Valsartan.

ELIGIBILITY:
Inclusion Criteria:

Patients hospitalized for COVID-19

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients with confirmed COVID-19 infection (any type), recruited in Italian hospital
Sampling Method: Non-Probability Sample
Enrollment: 3400 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Severe COVID-19 | 1 month
  Severity pneumonia or acute respiratory distress syndrome by COVID-19

SECONDARY OUTCOMES:
Death | 1 month
  Death by COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Di Castelnuovo, MSc, PhD, Principal Investigator — IRCCS Neuromed
Locations (1):
- IRCCS Neuromed, Department of Epidemiology and Prevention, Pozzilli, Italy

REFERENCES:
- [Derived] COVID-19 RISk and Treatments (CORIST) Collaboration. RAAS inhibitors are not associated with mortality in COVID-19 patients: Findings from an observational multicenter study in Italy and a meta-analysis of 19 studies. Vascul Pharmacol. 2020 Dec;135:106805. doi: 10.1016/j.vph.2020.106805. Epub 2020 Sep 28. PMID 32992048